CLINICAL TRIAL: NCT01761955
Title: Metabolic Health Benefits of Dairy Protein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: J2008:075
Record Dates: First submitted 2012-05-22; First posted 2013-01-07 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2008-12

CONDITIONS: Hyperlipidemia; Obesity
Keywords: body weight; lipids; glucose; insulin
MeSH Terms: conditions — Hyperlipidemias; Obesity; Body Weight; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dairy (Experimental): Consuming four or more servings of dairy per day.
  Interventions: Other: High Dairy
- Control, Low Dairy (Placebo Comparator): Participants consumed less than 2 servings of low fat dairy per day.

INTERVENTIONS:
Other: High Dairy — Consuming 4 or more servings of dairy products per day for a period of 6 months
  Arms: High Dairy

SUMMARY:
The purpose of this study is to evaluate the effects of regular low fat diary consumption on markers of cardiovascular (CV) and metabolic (cardiometabolic) health including body composition (% body fat, body weight), blood lipids, blood glucose, arterial compliance, blood pressure, insulin sensitivity and resting metabolic rate.

DETAILED DESCRIPTION:
This is a multi-centre, randomized, dietary intervention study of 12 months. A total of 100 overweight/obese individuals will be recruited, half recruited in Adelaide, South Australia and the other half from Manitoba, Canada. At baseline, subjects assigned to HD will be given standard serves of low fat dairy products (eg. 250mL milk, 200g yoghurt) on a regular basis for 6 months and asked to incorporate 4 serves/day into their diet. Volunteers randomized to the LD will be asked to continue with their habitual diet and consume less than 2 serves of dairy on a regular basis for 6 months. All participants will be asked to complete a food frequency questionnaire, physical activity diary, 3-day food record, and keep a record of dairy serves (food log) consumed each day. In total, participants will be asked to come to the centre 5 times throughout the study. However, the HD group will be asked to return to the centre every two weeks to receive diary product and return dairy record (food log). At baseline subjects will be asked to attend the Richardson Centre for Functional Foods and Nutraceuticals (RCFFN) fasted for various measurements including: body weight, blood pressure, arterial compliance, dual energy x-ray absorptiometry (DEXA) scan for measurement of body fat, abdominal fat and bone mineral density, waist and hip circumferences and provide a blood sample for the measurement of blood lipids, insulin and glucose.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25 kg/m2, assessed as age-related healthy based on pre-study screening examination including:

  * medical history
  * diet and lifestyle history
  * physical measurements (height, weight and blood pressure).

Exclusion Criteria:

* Pregnancy or likely to be pregnant (ionizing radiation from DEXA)
* Weight ≥135kg (exceeds the capacity of the DEXA scanner)diagnosed diabetes or cardiovascular disease
* Liver or renal disease
* Regular use of appetite suppressants
* Irregular use of other treatments which might interfere with the outcomes of the study (e.g anti-hypertensives, statins, thyroxine, omega-3 supplements etc).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
markers of metabolic (cardiometabolic) health | Six Months
  * total body composition (% body fat)
  * blood lipids, blood glucose
  * blood pressure
  * insulin sensitivity
  * resting metabolic rate

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Rempel, PhD, MBA, Principal Investigator — University of Manitoba; Gary Fulcher, PhD, Study Chair — University of Manitoba; Peter JH Jones, PhD, Study Director — University of Manitoba; Rotimi Aluko, PhD, Study Chair — University of Manitoba; Thomas Netticadan, PhD, Study Chair — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Rideout TC, Marinangeli CP, Martin H, Browne RW, Rempel CB. Consumption of low-fat dairy foods for 6 months improves insulin resistance without adversely affecting lipids or bodyweight in healthy adults: a randomized free-living cross-over study. Nutr J. 2013 May 2;12:56. doi: 10.1186/1475-2891-12-56. PMID 23638799